CLINICAL TRIAL: NCT06082765
Title: Cervical Cancer Screening with NGS-HPV Technology Based on Menstrual Blood
Status: Recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Collaborators: Wuhan Central Hospital (Other); Huanggang Maternal and Child Health Hospital (Unknown); Guilin People's Hospital (Unknown); Zaoyang Maternal and Child Health Hospital (Unknown); Jingshan People's Hospital (Unknown); Yichang Second People's Hospital (Other); Wuhan Third People's Hospital (Unknown); Dawu County People's Hospital (Unknown); Yingshan County People's Hospital (Unknown); Zhongxiang People's Hospital (Unknown); Zhongxiang Maternal and Child Health Hospital (Unknown); Wuxue First People's Hospital (Unknown); The First People's Hospital of Tianmen (Unknown); Huangmei County People's Hospital (Unknown); Huangmei Maternal and Child Health Care Hospital (Unknown); Gucheng County People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023071K
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: HPV; menstrual blood; cervical cancer; screening,
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The study aims to collect sanitary napkins for menstrual blood which contains cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our study is a population-based, cross-sectional study. This study is conducted to recruit cervical cancer screening participants to evaluate the application value of using high-throughput sequencing technology to detect HPV in menstrual blood for cervical cancer screening. Our study is designed as a two-phase study :

Phase I : This phase, which will be preparing to recruit 5,000 participants, evaluates the accuracy of menstrual blood (MB) self-sampling for detecting cervical intraepithelial neoplasia grade two or worse (CIN2+) in the general population, with a secondary objective to evaluate the Minipad as a special device to collect MB.

Phase II : This phase, which will continue to recruit toward the 10,000-participant target, will evaluate additional molecular markers (specifically DNA methylation) to optimize alternative triage methods for HPV-positive women in menstrual blood (MB) self-sampling. This phase aims to further reduce unnecessary colposcopies while maintaining high sensitivity for CIN2+ detection.

DETAILED DESCRIPTION:
Our study will recruit 10,000 participants for cervical cancer screening across seven sites in Hubei Province from September 1, 2023, to March 31, 2028. The participating sites include: Fruit Lake Community (where Zhongnan Hospital of Wuhan University is located), Jiang'an District (Wuhan Central Hospital), Huangzhou district of Huanggang County (Huanggang Maternal and Child Health Care Hospital), Jingling Community of Tianmen County (the First People's Hospital of Tianmen), Liutang Community of Huangmei County (Huangmei County People's Hospital), Gongtang Community of Zhongxiang City (Zhongxiang Maternal and Child Health Care Hospital), and Chaihu Community of Zhongxiang City (People's Hospital of Zhongxiang).. The procedures were conducted as below: (1) Conduct cervical cancer screening (TCT+hr-HPV) for all the participants. (2) Collect sanitary napkins from participants during their first menstrual period after cervical HPV testing. (3) Detect HPV using high-throughput sequencing technology in the menstrual blood (MB) from sanitary napkins. (4) Colposcopy referral (biopsy if necessary) for patients with abnormal screening results. (5) Compare the concordance between MB-HPV and clinician-collected HPV. (6) Evaluate the accuracy of menstrual blood (MB) self-sampling for detecting cervical intraepithelial neoplasia grade two or worse (CIN2+) in the general population, with a secondary objective to evaluate the Minipad as a special device to collect MB. (7) Evaluate additional molecular markers (specifically DNA methylation) to optimize alternative triage methods for HPV-positive women in menstrual blood (MB) self-sampling.

ELIGIBILITY:
Inclusion Criteria:

1. plan to undergo cervical screening
2. with regular menstruation (21-35 days)
3. agree to participate in this study and have signed an informed consent form

Exclusion Criteria:

1. with amenorrhea or menopause
2. suffering from genital tract infection
3. refuse to participate in this study

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our study is designed as a two-phase study. The phase I aims to recruit 5,000 women to explore the application value of HPV detection in menstrual blood using next-generation sequencing. The phase II aims to recruit 5,000 women to evaluate additional molecular markers (specifically DNA methylation) to optimize alternative triage methods for HPV-positive women in menstrual blood (MB) self-sampling.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
HPV detection in menstrual blood | December 31, 2025
  In phase I: The primary aim of this study is to evaluate the accuracy of menstrual blood (MB) self-sampling for detecting cervical intraepithelial neoplasia grade two or worse (CIN2+) in the general population.
  In phase II: The primary aim of this study is to evaluate additional molecular markers (specifically DNA methylation) to optimizeThis phase, which will continue to recruit toward the 10,000-participant target, will evaluate additional molecular markers (specifically DNA methylation) to optimize alternative triage methods for HPV-positive women in menstrual blood (MB) self-sampling.

SECONDARY OUTCOMES:
HPV detection in menstrual blood | December 31, 2025
  The secondary objective of this study is to evaluate the accuracy of minipad as a special device for menstrual blood (MB) collection in detecting grade 2 or more cervical intraepithelial neoplasia (CIN2+) in the general population

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Hu, doctor, Principal Investigator — Zhongnan Hospital
Locations (1):
- Department of Gynecologic Oncology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Tian X, Cao C, Wang L, Zhang J, Chen Y, Tian R, Zhou B, Sun L, Zhang C, Gan L, Jin Y, Liu J, Wang T, Shen Y, Huang S, Zhang L, Zhang S, Chen P, Tong C, Kang J, Fan H, Zhou G, Xiang L, Wen Y, Gan R, Chen Y, Li X, Zhai L, Zhang Q, Ma D, Han Z, Hu Z. Testing menstrual blood for human papillomavirus during cervical cancer screening in China: cross sectional population based study. BMJ. 2026 Feb 4;392:e084831. doi: 10.1136/bmj-2025-084831. PMID 41638692